CLINICAL TRIAL: NCT04969276
Title: A Phase II, Open-label Study to Assess the Safety and Immunogenicity of Fluzone® High-Dose Quadrivalent (Influenza Vaccine), 2021-2022 Formulation and a Third Dose of Moderna COVID-19 Vaccine (mRNA-1273 Vaccine) Administered Either Concomitantly or Singly in Adults 65 Years of Age and Older Previously Vaccinated With a 2-dose Schedule of Moderna COVID-19 Vaccine
Brief Title: Study of a Quadrivalent High-Dose Influenza Vaccine and a Moderna COVID-19 Vaccine Administered Either Concomitantly or Singly in Participants 65 Years of Age and Older Previously Vaccinated With a 2-dose Schedule of Moderna COVID-19 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QHD00028; U1111-1266-7472 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-07-16; First posted 2021-07-20 (Actual); Results first posted 2022-12-13 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Influenza Immunization; Healthy Volunteers
MeSH Terms: conditions — Influenza, Human | interventions — CVnCoV COVID-19 vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: Fluzone High-Dose (HD) Quadrivalent Influenza Vaccine and COVID-19 Vaccine (Experimental): Participants received an injection of 0.7 milliliters (mL), fluzone HD quadrivalent influenza vaccine, co-administered with 0.5 mL COVID-19 vaccine, intramuscularly (IM) on Day 1.
  Interventions: Biological: Quadrivalent Inactivated Influenza High Dose; Biological: COVID-19 mRNA Vaccine (nucleoside modified)
- Group 2: Fluzone HD Quadrivalent Influenza Vaccine (Active Comparator): Participants received a single injection of 0.7 mL fluzone HD quadrivalent influenza vaccine, IM on Day 1.
  Interventions: Biological: Quadrivalent Inactivated Influenza High Dose
- Group 3: COVID-19 Vaccine (Active Comparator): Participants received a single injection of 0.5 mL COVID-19 mRNA Vaccine, IM on Day 1.
  Interventions: Biological: COVID-19 mRNA Vaccine (nucleoside modified)

INTERVENTIONS:
Biological: Quadrivalent Inactivated Influenza High Dose — Sterile suspension for injection in a pre-filled syringe Intramuscular injection
  Other Names: Fluzone HD Quadrivalent vaccine
  Arms: Group 1: Fluzone High-Dose (HD) Quadrivalent Influenza Vaccine and COVID-19 Vaccine; Group 2: Fluzone HD Quadrivalent Influenza Vaccine
Biological: COVID-19 mRNA Vaccine (nucleoside modified) — Sterile suspension (white to off-white) in multidose vial Intramuscular injection
  Other Names: Moderna COVID-19 Vaccine (mRNA-1273 vaccine)
  Arms: Group 1: Fluzone High-Dose (HD) Quadrivalent Influenza Vaccine and COVID-19 Vaccine; Group 3: COVID-19 Vaccine

SUMMARY:
The main purpose of this Phase II study was to assess the safety and immunogenicity of a dose of Fluzone High-Dose (HD) Quadrivalent vaccine and a third dose or booster dose of Moderna coronavirus disease 19 (COVID-19) vaccine administered concomitantly or singly in adults 65 years of age and older having received their second dose of the 2-dose schedule of Moderna COVID-19 vaccine at least 5 months before enrollment in the study.

DETAILED DESCRIPTION:
Participants were in the study for 6 months (approximately 180 days).

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to >= 65 years of age on the day of inclusion.
* In good health or with underlying medical condition(s) that were judged to be stable by the Investigator. A stable medical condition was defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
* Participants who previously received 2 injections of Moderna COVID-19 Vaccine with the second dose received at least 5 months before Visit 1.
* Abled to attend all scheduled visits and to complied with all study procedures.

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the 3 months preceding planned inclusion).
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances.
* Previous dermal filler injection (either lips or face fillers).
* Thrombocytopenia, contraindicated IM injection.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicated IM vaccination.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of study intervention administration or febrile illness (temperature >= 100.4°Fahrenheit [F] [38.0° Celsius {C}]). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* History of serious adverse reaction to any influenza or COVID-19 vaccines.
* Personal history of Guillain-Barré syndrome (GBS).
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.
* Any condition that in the opinion of the Investigator posed a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine.
* Receipt of any vaccine in the 4 weeks preceding the study intervention(s) administration or planned receipt of any vaccine in the period between Visit 01 and 4 weeks following the study intervention(s) administration. Note: Vaccination of Group 3 participants with Fluzone High-Dose Quadrivalent vaccine at the end of the study was not considered by the Sponsor as meeting this exclusion criterion.
* Receipt of blood-derived immune globulins, blood, or blood-derived products in the past 3 months.
* Participation at the time of study enrollment (or in the 30 days preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating vaccine, drug, medical device, or medical procedure.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 306 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- United States (6):
  - Investigational Site Number :8400003, Glendale, Arizona
  - Investigational Site Number :8400006, San Diego, California
  - Investigational Site Number :8400004, Vista, California
  - Investigational Site Number :8400005, Centennial, Colorado
  - Investigational Site Number :8400001, Peoria, Illinois
  - Investigational Site Number :8400002, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Izikson R, Brune D, Bolduc JS, Bourron P, Fournier M, Moore TM, Pandey A, Perez L, Sater N, Shrestha A, Wague S, Samson SI. Safety and immunogenicity of a high-dose quadrivalent influenza vaccine administered concomitantly with a third dose of the mRNA-1273 SARS-CoV-2 vaccine in adults aged >/=65 years: a phase 2, randomised, open-label study. Lancet Respir Med. 2022 Apr;10(4):392-402. doi: 10.1016/S2213-2600(21)00557-9. Epub 2022 Feb 1. PMID 35114141
- See also: QHD00028 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25343&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 sites in the United States. A total of 306 participants were enrolled between 16 July 2021 to 05 August 2021.
Pre-assignment Details: A total of 296 participants were vaccinated in the study.
Period: Overall Study
Arm/Group | Group 1: Fluzone High-Dose (HD) Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Started | 100 | 101 | 105
Safety Analysis Set (SafAS) (SafAS included all participants who had received the study vaccine(s) and were analyzed according to the vaccine they actually received and study intervention group.) | 100 | 92 | 104
Completed | 99 | 89 | 105
Not Completed | 1 | 12 | 0
Not completed — Protocol Deviation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 10 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine: Participants received an injection of 0.7 mL, fluzone HD quadrivalent influenza vaccine, co-administered with 0.5 mL COVID-19 vaccine, IM on Day 1.
- Total: Total of all reporting groups
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine | Total
Number analyzed (Participants) | 100 | 101 | 105 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (4.76) | 71.7 (5.16) | 72.0 (4.89) | 71.7 (4.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 63 | 172
  Male | 45 | 47 | 42 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 3
  Black or African American | 1 | 4 | 0 | 5
  White | 94 | 95 | 103 | 292
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report form (CRF) in terms of diagnosis and onset window post-vaccination. All participants were observed for 30 minutes after vaccination, and any unsolicited AEs that occurred during that time were recorded as immediate unsolicited AEs in the CRF. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 30 minutes post vaccination
Population: Analysis was performed on SafAS which included all participants who had received the study vaccine(s) and were analyzed according to the vaccine they actually received and study intervention group.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 100 | 92 | 104
Participants | 1 | 1 | 0

2. Primary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction (SR) was an "expected" adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF. Solicited injection site reactions included injection site pain, axillary swelling and tenderness, injection site erythema, injection site swelling, injection site induration, and injection site bruising. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 7 days post-vaccination
Population: Analysis was performed on the SafAS. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 100 | 89 | 104
Participants
  Injection site pain | 82 | 54 | 92
  Axillary swelling | 2 | 2 | 1
  Axillary tenderness | 3 | 3 | 3
  Injection site erythema | 22 | 10 | 32
  Injection site swelling | 15 | 6 | 27
  Injection site induration | 12 | 3 | 22
  Injection site bruising | 7 | 0 | 4

3. Primary Outcome: Number of Participants With Solicited Systemic Reactions
Description: A SR was an "expected" adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the protocol and CRF. Solicited systemic reactions included fever, headache, malaise, myalgia, arthralgia, shivering, fatigue, nausea and vomiting. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 7 days post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 100 | 89 | 104
Participants
  Fever | 12 | 1 | 12
  Headache | 52 | 18 | 55
  Malaise | 46 | 13 | 59
  Myalgia | 50 | 20 | 64
  Arthralgia | 24 | 8 | 27
  Shivering | 32 | 6 | 22
  Fatigue | 62 | 26 | 73
  Nausea | 32 | 5 | 27
  Vomiting | 4 | 3 | 1

4. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRF in terms of diagnosis and/or onset window post-vaccination. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 21 days post-vaccination
Population: Analysis was performed on the SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 100 | 92 | 104
Participants | 17 | 11 | 15

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Event of Special Interest (AESIs)
Description: An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. AESIs was defined as one of scientific and medical concern specific to the sponsor's study intervention or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor was done. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: From Day 1 up to 6 months post-vaccination
Population: Analysis was performed on the SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 100 | 92 | 104
Participants
  SAEs | 2 | 0 | 3
  AESIs | 1 | 0 | 1

6. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs)
Description: A MAAE was a new onset or a worsening of a condition that prompted the participant or participant's parent/legally acceptable representative to seek unplanned medical advice at a physician's office or emergency department including medical advice seeking during the study visit or routine medical care. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: From Day 1 up to 6 months post-vaccination
Population: Analysis was performed on the SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 100 | 92 | 104
Participants | 10 | 6 | 17

7. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine and COVID-19 Vaccine Antibodies at Day 1
Description: GMTs of anti-influenza and anti-COVID-19 antibodies were measured using hemagglutination inhibition (HAI) assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Yamagata, and B/Victoria. Titers were expressed in terms of 1/dilution.
Time Frame: Day 1 (pre-vaccination)
Population: Analysis was performed on Immunogenicity analysis set which included all randomized participants who received at least 1 dose of the study vaccine and analyzed according to the vaccine they actually received and study intervention group. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 99 | 91 | 101
titers
  A/H1N1: Pre-vaccination | 55.8 [44.2 to 70.4] | 45.5 [34.7 to 59.7] | 49.7 [37.7 to 65.4]
  A/H3N2: Pre-vaccination | 95.0 [77.5 to 116] | 85.4 [66.3 to 110] | 80.3 [63.1 to 102]
  B/Yamagata: Pre-vaccination | 221 [178 to 274] | 204 [159 to 262] | 203 [163 to 252]
  B/Victoria: Pre-vaccination | 163 [137 to 194] | 155 [127 to 190] | 165 [136 to 201]

8. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine and COVID-19 Vaccine Antibodies at Day 22
Description: GMTs of anti-influenza and anti-COVID-19 antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Yamagata, and B/Victoria. Titers were expressed in terms of 1/dilution.
Time Frame: Day 22 (post-vaccination)
Population: Analysis was performed on Immunogenicity analysis set. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 97 | 86 | 102
titers
  A/H1N1: Post-vaccination | 363 [276 to 476] | 366 [272 to 491] | 41.2 [31.4 to 54.2]
  A/H3N2: Post-vaccination | 286 [233 to 352] | 315 [257 to 386] | 76.5 [61.1 to 95.8]
  B/Yamagata: Post-vaccination | 429 [350 to 525] | 471 [378 to 588] | 198 [160 to 243]
  B/Victoria: Post-vaccination | 377 [325 to 438] | 390 [327 to 465] | 176 [146 to 212]

9. Primary Outcome: Geometric Mean Titers Ratio (GMTR) of Influenza Vaccine and COVID-19 Vaccine Antibodies
Description: GMTs of anti-influenza and anti-COVID-19 antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. GMTRs were calculated as the ratio of GMTs post-vaccination (on Day 22) and pre-vaccination (on Day 1) i.e., Day 22/Day 01.
Time Frame: Day 1 (pre-vaccination) and Day 22 (post-vaccination)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 96 | 86 | 100
ratio
  A/H1N1 | 6.35 [4.88 to 8.26] | 8.10 [6.09 to 10.8] | 0.868 [0.821 to 0.917]
  A/H3N2 | 3.06 [2.54 to 3.70] | 3.54 [2.82 to 4.45] | 0.940 [0.870 to 1.01]
  B/Yamagata | 1.94 [1.68 to 2.23] | 2.27 [1.84 to 2.79] | 0.983 [0.918 to 1.05]
  B/Victoria | 2.27 [1.96 to 2.63] | 2.44 [2.01 to 2.96] | 1.05 [0.972 to 1.14]

10. Primary Outcome: Percentage of Participants With Antibody Titers Greater Than or Equal to (>=)10 (1/Dilution)
Description: Anti-influenza and anti-COVID 19 antibodies were measured using HAI assay method for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. Percentage of participants with HAI titers >=10 (1/dilution) are reported in the outcome measure.
Time Frame: Day 1 (pre-vaccination)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 99 | 91 | 101
percentage of participants
  A/H1N1: Pre-vaccination | 97.0 [91.4 to 99.4] | 94.5 [87.6 to 98.2] | 91.1 [83.8 to 95.8]
  A/H3N2: Pre-vaccination | 100 [96.3 to 100] | 98.9 [94.0 to 100] | 99.0 [94.6 to 100]
  B/Yamagata: Pre-vaccination | 100 [96.3 to 100] | 100 [96.0 to 100] | 99.0 [94.6 to 100]
  B/Victoria: Pre-vaccination | 100 [96.3 to 100] | 100 [96.0 to 100] | 100 [96.4 to 100]

11. Primary Outcome: Percentage of Participants With Antibody Titers Greater Than or Equal to (>=)10 (1/Dilution)
Description: as for outcome 10
Time Frame: Day 22 (post-vaccination)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 97 | 86 | 102
percentage of participants
  A/H1N1: Post-vaccination | 100 [96.3 to 100] | 100 [95.8 to 100] | 91.2 [83.9 to 95.9]
  A/H3N2: Post-vaccination | 100 [96.3 to 100] | 100 [95.8 to 100] | 99.0 [94.7 to 100]
  B/Yamagata: Post-vaccination | 100 [96.3 to 100] | 100 [95.8 to 100] | 99.0 [94.7 to 100]
  B/Victoria: Post-vaccination | 100 [96.3 to 100] | 100 [95.8 to 100] | 100 [96.4 to 100]

12. Primary Outcome: Percentage of Participants Achieving Seroconversion Against Influenza and COVID-19 Virus Antigens
Description: Anti-influenza and anti-COVID-19 antibodies were measured by HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. Seroconversion was defined as either a pre-vaccination HAI titer less than (<)10 (1/dilution) and a post-vaccination titer >=40 (1/dilution) or a pre-vaccination titer >=10 (1/dilution) and a >= four-fold increase in post-vaccination titer at Day 22.
Time Frame: Day 22 (post-vaccination)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 96 | 86 | 100
percentage of participants
  A/H1N1 | 68.8 [58.5 to 77.8] | 72.1 [61.4 to 81.2] | 0.0 [0.0 to 3.6]
  A/H3N2 | 43.8 [33.6 to 54.3] | 47.7 [36.8 to 58.7] | 0.0 [0.0 to 3.6]
  B/Yamagata | 17.7 [10.7 to 26.8] | 20.9 [12.9 to 31.0] | 1.0 [0.0 to 5.4]
  B/Victoria | 30.2 [21.3 to 40.4] | 24.4 [15.8 to 34.9] | 1.0 [0.0 to 5.4]

13. Primary Outcome: Percentage of Participants With Antibody Titers >=40 (1/Dilution)
Description: Anti-influenza and anti-COVID 19 antibodies were measured using HAI assay method for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. Percentage of participants with HAI titers >=40 (1/dilution) are reported in the outcome measure.
Time Frame: Day 1 (pre-vaccination)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 99 | 91 | 101
percentage of participants
  A/H1N1: Pre-vaccination | 65.7 [55.4 to 74.9] | 56.0 [45.2 to 66.4] | 59.4 [49.2 to 69.1]
  A/H3N2: Pre-vaccination | 83.8 [75.1 to 90.5] | 79.1 [69.3 to 86.9] | 77.2 [67.8 to 85.0]
  B/Yamagata: Pre-vaccination | 97.0 [91.4 to 99.4] | 90.1 [82.1 to 95.4] | 96.0 [90.2 to 98.9]
  B/Victoria: Pre-vaccination | 99.0 [94.5 to 100] | 94.5 [87.6 to 98.2] | 95.0 [88.8 to 98.4]

14. Primary Outcome: Percentage of Participants With Antibody Titers >=40 (1/Dilution)
Description: as for outcome 13
Time Frame: Day 22 (post-vaccination)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 97 | 86 | 102
percentage of participants
  A/H1N1: Post-vaccination | 94.8 [88.4 to 98.3] | 95.3 [88.5 to 98.7] | 53.9 [43.8 to 63.8]
  A/H3N2: Post-vaccination | 96.9 [91.2 to 99.4] | 100 [95.8 to 100] | 72.5 [62.8 to 80.9]
  B/Yamagata: Post-vaccination | 100 [96.3 to 100] | 98.8 [93.7 to 100] | 96.1 [90.3 to 98.9]
  B/Victoria: Post-vaccination | 100 [96.3 to 100] | 100 [95.8 to 100] | 96.1 [90.3 to 98.9]

15. Primary Outcome: Geometric Mean Concentration (GMC) of Anti-S Binding Immunoglobulin G (IgG) Antibodies
Description: GMCs of Anti-S binding IgG antibodies were assessed using enzyme-linked immunosorbent assay (ELISA) method and were measured in binding antibody units/milliliter (BAU/mL).
Time Frame: Day 1 (pre-vaccination)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: BAU/mL
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 99 | 91 | 102
BAU/mL | 565 [479 to 666] | 462 [382 to 560] | 552 [461 to 662]

16. Primary Outcome: Geometric Mean Concentration (GMC) of Anti-S Binding Immunoglobulin G (IgG) Antibodies
Description: GMCs of Anti-S binding IgG antibodies were assessed using ELISA method and were measured in BAU/mL.
Time Frame: Day 22 (post-vaccination)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: BAU/mL
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 97 | 86 | 103
BAU/mL | 7634 [6445 to 9042] | 395 [311 to 502] | 7904 [6883 to 9077]

17. Primary Outcome: Geometric Mean Concentration Ratio (GMCR) of Anti-S Binding IgG Antibodies
Description: GMCs of Anti-S binding IgG antibodies were assessed using ELISA method. GMCR was calculated as the ratio of GMC post-vaccination (on Day 22) and pre-vaccination (on Day 1) i.e., Day 22/Day 01.
Time Frame: Day 1 (pre-vaccination) and Day 22 (post-vaccination)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 96 | 86 | 102
ratio | 13.7 [11.2 to 16.8] | 0.875 [0.745 to 1.03] | 14.2 [12.0 to 16.9]

18. Primary Outcome: Percentage of Participants With >=2-Fold and >=4-Fold Rise in Anti-S Binding IgG Antibodies
Description: Percentage of participants with >=2-fold and >=4-fold rise in Anti-S binding IgG antibodies at Day 22 (post-vaccination) are reported in this outcome measure. Percentage of participants with >=2-fold rise are those for whom the computed value at Day 22 was *2 compared to the computed value at Day 1 and percentage of participants with >=4-fold rise are those for whom the computed value at Day 22 was *4 compared to the computed value at Day 1.
Time Frame: Day 22 (post-vaccination)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Fluzone HD Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
Number analyzed (Participants) | 96 | 86 | 102
percentage of participants
  >= 2-fold rise | 97.9 [92.7 to 99.7] | 3.5 [0.7 to 9.9] | 98.0 [93.1 to 99.8]
  >= 4-fold rise | 92.7 [85.6 to 97.0] | 2.3 [0.3 to 8.1] | 95.1 [88.9 to 98.4]

ADVERSE EVENTS:
Time Frame: Unsolicited AEs were collected from Day 1 up to 21 days post-vaccination. SR data were collected up to 7 days post-vaccination. SAE data were collected from Day 1 up to 6 months post-vaccination
Description: SR: "expected" adverse reaction (sign/symptom) observed & reported under conditions (nature and onset) prelisted (i.e., solicited) in protocol and CRF & considered as related to IMP administered. Unsolicited AE: AE that did not fulfill conditions prelisted (i.e., solicited) in CRF in terms of diagnosis & onset window post-vaccination. SafAS. In AE section, SR Fever & shivering are reported as Pyrexia & chills respectively. Reported AEs for each arm were presented as pre-specified in protocol.
Groups:
- Group 1: Fluzone High-Dose (HD) Quadrivalent Influenza Vaccine and COVID-19 Vaccine: Participants received an injection of 0.7 mL, fluzone HD quadrivalent influenza vaccine, co-administered with 0.5 mL COVID-19 vaccine, IM on Day 1.
Arm/Group | Group 1: Fluzone High-Dose (HD) Quadrivalent Influenza Vaccine and COVID-19 Vaccine | Group 2: Fluzone HD Quadrivalent Influenza Vaccine | Group 3: COVID-19 Vaccine
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/92 | 0/104
Serious Adverse Events (participants affected / at risk) | 2/100 | 0/92 | 3/104
Other Adverse Events (participants affected / at risk) | 94/100 | 65/92 | 100/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Fluzone High-Dose (HD) Quadrivalent Influenza Vaccine and COVID-19 Vaccine (N=100) | Group 2: Fluzone HD Quadrivalent Influenza Vaccine (N=92) | Group 3: COVID-19 Vaccine (N=104)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid Mass (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Fluzone High-Dose (HD) Quadrivalent Influenza Vaccine and COVID-19 Vaccine (N=100) | Group 2: Fluzone HD Quadrivalent Influenza Vaccine (N=92) | Group 3: COVID-19 Vaccine (N=104)
Nausea (Gastrointestinal disorders) | 32 (32) | 6 (6) | 27 (27) — Nausea events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Chills (General disorders) | 32 (32) | 6 (6) | 22 (22)
Fatigue (General disorders) | 62 (62) | 26 (26) | 73 (73)
Injection Site Bruising (General disorders) | 7 (8) | 0 (0) | 4 (4)
Injection Site Erythema (General disorders) | 22 (28) | 10 (10) | 32 (32)
Injection Site Induration (General disorders) | 12 (12) | 3 (3) | 22 (22)
Injection Site Pain (General disorders) | 82 (139) | 54 (54) | 92 (92)
Injection Site Swelling (General disorders) | 15 (17) | 6 (6) | 27 (27)
Malaise (General disorders) | 46 (46) | 13 (13) | 59 (59)
Pyrexia (General disorders) | 12 (12) | 1 (1) | 13 (13) — Pyrexia/Fever events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (24) | 8 (8) | 27 (28)
Myalgia (Musculoskeletal and connective tissue disorders) | 50 (50) | 20 (20) | 64 (64)
Headache (Nervous system disorders) | 52 (52) | 18 (18) | 55 (55)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT04969276/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT04969276/SAP_001.pdf